CLINICAL TRIAL: NCT00198393
Title: Randomized Phase 2 Study of 3 Therapeutic Modalities in PS 2/3 Patients With NSCLC Stage IIIB/IV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Collaborators: AstraZeneca (Industry); Sanofi (Industry)
Responsible Party: Pr Jean-François Morère, Intergroupe Francophone de Cancérologie Thoracique
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-0301
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2010-04-30 (Estimated); Status verified 2010-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: stage IIIB/IV NSCLC; patients with performance status 2 or 3.
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Gefitinib
  Interventions: Drug: Gefitinib
- B (Experimental): Gemcitabine
  Interventions: Drug: gemcitabine
- C (Experimental): Docetaxel
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Gefitinib — 250 mg/day, until progression
  Arms: A
Drug: gemcitabine — 1250 mg/m² D1 and D8 (D1=D28, until progression)
  Arms: B
Drug: Docetaxel — 75 mg/m² D1 (D1=D22, until progression)
  Arms: C

SUMMARY:
Patients presenting a deterioration of the general state (performance status [PS] 2-3), constitute a population which needs an adapted treatment. An analysis was made of the evolution of PS 2 patients included in the Eastern Cooperative Oncology Group (ECOG) 1594 trial which evaluated associations of new cytotoxic agents (gemcitabine, paclitaxel, docetaxel) with cisplatin. During this trial, the inclusion of these patients stopped due to the occurrence of toxicities more frequent than in the other populations (PS 0-1). At the end of this study, with the analysis of total toxicity, this one was not higher than that noted in the groups of PS 0 and 1 patients. In the population of PS 2 patients, 5 deaths had been noted, but the analysis showed that only 2 were due to the treatment. It was noted that the lower survival compared to the others was related to the disease and not to the treatment. These patients are often symptomatic and need palliative treatment. The benefit of chemotherapy should not be denied. They should profit from a monochemotherapy with the new cytotoxic agents, without associated platinum salt.

DETAILED DESCRIPTION:
Arm A Iressa 250 mg daily PROG/TOX --> Taxotere 75 mg/m² d1 (d1=d22)

Arm B Gemzar 1250 mg/m² d1 & d8 (d1=d22) PROG/TOX --> Iressa 250 mg daily

Arm C Taxotere 75 mg/m² d1 (d1=d22) PROG/TOX --> Iressa 250 mg daily

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIB/IV NSCLC
* patients with performance status 2 or 3.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2004-11; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | week

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Morere, Pr, Principal Investigator — Intergroupe Francophone de Cancerologie Thoracique; Denis Moro-Sibilot, Pr, Principal Investigator — Intergroupe Francophone de Cancerologie Thoracique
Locations (2):
- France (2):
  - CHU Avicenne - Oncologie, Bobigny
  - CHU Grenoble - pneumologie, Grenoble

REFERENCES:
- [Background] Moro-Sibilot D, Pluquet E, Zalcman G, Brechot JM, Souquet PJ, Debieuvre D, Morin F, Morere JF. [What treatment for a patient of PS 2-3 with stage IV non-small cell lung cancer?]. Rev Mal Respir. 2007 Oct;24(8 Pt 2):6S120-4. French. PMID 18235404
- [Result] Morere JF, Brechot JM, Westeel V, Gounant V, Lebeau B, Vaylet F, Barlesi F, Urban T, Souquet PJ, Debieuvre D, Baudrin L, Zalcman G, Morin F, Milleron B, Moro-Sibilot D. Randomized phase II trial of gefitinib or gemcitabine or docetaxel chemotherapy in patients with advanced non-small-cell lung cancer and a performance status of 2 or 3 (IFCT-0301 study). Lung Cancer. 2010 Dec;70(3):301-7. doi: 10.1016/j.lungcan.2010.03.003. Epub 2010 Apr 18. PMID 20400201
- See also: Official website — http://www.ifct.fr